CLINICAL TRIAL: NCT05931380
Title: A Phase 3, Randomized, Double-Blind Study to Investigate the Efficacy and Safety of Once-Daily Oral LY3502970 Compared With Placebo in Japanese Adult Participants With Obesity Disease
Brief Title: A Study of Once-Daily Oral Orforglipron (LY3502970) in Japanese Adult Participants With Obesity Disease
Acronym: ATTAIN-J
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18744; J2A-JE-GZPD (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-06-27; First posted 2023-07-05 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: Overweight; Metabolism and Nutrition Disorder
MeSH Terms: conditions — Obesity; Overweight; Nutrition Disorders | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Orforglipron Dose 1 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 2 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 3 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Arms: Orforglipron Dose 1; Orforglipron Dose 2; Orforglipron Dose 3
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to investigate the efficacy and safety of oral orforglipron in participants with obesity disease with obesity-related health problems.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a BMI ≥27 kg/m² and <35 kg/m² and at least 2 obesity-related health problems (treated or untreated), OR a BMI ≥35 kg/m² and at least 1 obesity-related health problem (treated or untreated). At least one obesity-related health problem should be hypertension, dyslipidemia or T2D (approximately 25% of participants).
* Have a history of at least one self-reported unsuccessful dietary effort to lose body weight.
* Males and females may participate in this trial. Female participants must not be pregnant, intending to be pregnant, breastfeeding, or intending to breastfeed.
* Contraceptive use by participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* No male contraception is required except in compliance with specific local government study requirements.

Exclusion Criteria:

* For participants with Type 2 Diabetes (T2D):

  * Have Type 1 Diabetes (T1D), history of ketoacidosis or hyperosmolar state/coma, or any other types of diabetes except T2D.
  * Have had 1 or more episode of severe hypoglycemia and/or 1 or more episode of hypoglycemia unawareness within the 180 days prior to screening.
* Have renal impairment measured as estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m², calculated by Japanese Society of Nephrology coefficient-modified chronic kidney disease-epidemiology equation during screening.
* Have a known clinically significant gastric emptying abnormality.
* For participants without Type 2 diabetes (T2D): Have any type of diabetes with hemoglobin A1c (HbA1c) ≥6.5 %.
* Have a self-reported change in body weight >5 kg (11 pounds) within 90 days prior to screening.
* Have chronic kidney disease.
* Have lupus or rheumatoid arthritis.
* Have the following cardiovascular conditions within 90 days prior to screening.
* Have acute or chronic hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Mean Percent Change in Body Weight | Baseline, Week 72
Percentage of Participants Who Achieve ≥5% Body Weight Reduction | Baseline to Week 72

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve ≥10% Body Weight Reduction | Baseline to Week 72
Percentage of Participants Who Achieve ≥15% Body Weight Reduction | Baseline to Week 72
Percentage of Participants Who Achieve ≥20% Body Weight Reduction | Baseline to Week 72
Mean Change from Baseline in Body Mass Index (BMI) | Baseline, Week 72
Percentage of Participants Who Had Improvements in Hypertension | Baseline to Week 72
Percentage of Participants Who Had Improvements in Dyslipidemia (only for participants with Dyslipidemia at baseline) | Baseline to Week 72
Percentage of Participants Who Achieve HbA1c Target value (<6.5% (48 mmol/mol) at Week 72 (only T2D at Baseline): | Baseline to Week 72
Mean Change from Baseline in Visceral Adipose Tissue (VAT) | Baseline, Week 72
Mean Change from Baseline in Waist Circumference at Umbilical Level | Baseline, Week 72
Mean Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 72
Mean Change from Baseline in non-High Density Lipoprotein (HDL) | Baseline, Week 72
Mean Change from Baseline in HDL | Baseline, Week 72
Mean Change from Baseline in Triglycerides | Baseline, Week 72
Mean Change from Baseline in Fasting Glucose | Baseline, Week 72
Mean Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 72
Mean Change from Baseline in High-sensitivity C-reactive Protein | Baseline, Week 72
Mean Change from Baseline in Short Form 36 Version 2 (SF-36v2) Acute Form Domain Scores | Baseline, Week 72
Mean Change from Baseline in IMPACT of Weight on Quality-of-Life Lite Clinical Trials Version (IWQOL-Lite-CT) Physical Function, Physical, and Psychosocial Composite Score | Baseline, Week 72
Time to Onset of Type 2 Diabetes (T2D) (only non T2D at Baseline) | Baseline to Week 72
Pharmacokinetics (PK): Plasma Concentration of Orforglipron | Baseline to Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- Japan (16):
  - Nishiyamadou Keiwa Hospital, Naka, Ibaraki
  - Tsuchiura Beryl Clinic, Tsuchiura, Ibaraki
  - Ohishi Internal Medicine Clinic, Tsuchiura, Ibaraki
  - Shonan Takai Clinic, Kamakura, Kanagawa
  - Takai Internal Medicine Clinic, Kamakura-shi, Kanagawa
  - Medical Corporation Yuga Higashirinkan Kaneshiro Diabetes Clinic, Sagamihara, Kanagawa
  - Shiraiwa Medical Clinic, Kashihara, Osaka
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Sugiura Clinic, Kawaguchi, Saitama
  - Yotsuya Medical Cube, Chiyoda City, Tokyo
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Heishinkai Medical Group ToCROM Clinic, Shinjuku-ku, Tokyo
  - Hiroshima Station Clinic, Hiroshima
  - Osaka Nishiumeda Clinic, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/